CLINICAL TRIAL: NCT06206824
Title: Randomized, Double-Blind, Placebo-Controlled Phase 1 Study to Evaluate Safety, Tolerability, PK/PD of SAD, MAD and Food Effect of Leucettinib-21 in Healthy Male Subjects, and Single Dose in Subjects With Down Syndrome or Alzheimer's Disease
Brief Title: Leucettinib-21 First-in-Human Phase 1 in Healthy Volunteers and Subjects With Down Syndrome and Alzheimer's Disease
Acronym: LEUCETTA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Perha Pharmaceuticals (Industry)
Collaborators: France 2030 program (Unknown); European Innovation Council (Other); Fondation Jérôme Lejeune (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP112522; 2023-507075-22 (EudraCT Number)
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Down Syndrome; Alzheimer's Disease
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 : Single Ascending Doses in Healthy Volunteers (Experimental): A total of 48 healthy male volunteers will be randomized into six consecutive single ascending dose cohorts of 8 subjects, 6 receiving one dose of Leucettinib-21 and 2 receiving placebo.
  Interventions: Drug: Leucettinib-21
- Part 2 : Food-Effect in Healthy Volunteers (Experimental): A total of 12 healthy male volunteers will be randomly assigned to one of two sequences in this cross over study part. All subjects will receive the same one dose of Leucettinib-21 in each sequence.
  Interventions: Drug: Leucettinib-21
- Part 3 : Multiple Ascending Doses over 14 days in Healthy Volunteers (Experimental): A total of 36 healthy male volunteers will be randomized into three consecutive multiple ascending doses cohorts of 12 subjects, 9 receiving one dose of Leucettinib-21 and 3 receiving placebo everyday for 14 days.
  Interventions: Drug: Leucettinib-21
- Part 4 : Single Dose in People with Down Syndrome and Alzheimer's Disease (Experimental): A total of 12 people with Down Syndrome and 12 people with Alzheimer's Disease will receive the same one dose of Leucettinib-21.
  Interventions: Drug: Leucettinib-21
- Part 5 : Single Ascending Doses in Healthy Volunteers (Experimental): A total of 32 healthy volunteers will be randomized into three consecutive single ascending dose cohorts, of 16 male and female subjects for the first cohort, 12 receiving one dose of Leucettinib-21 and 4 receiving placebo, and 8 male subjects for the two following cohorts, 6 receiving one dose of Leucettinib-21 and 2 receiving placebo.
  Interventions: Drug: Leucettinib-21
- Part 6 : Single dose over 14 days in Healthy Volunteers (Experimental): A total of 12 healthy male volunteers will be randomized into one cohort of 12 subjects, 9 receiving one dose of Leucettinib-21 and 3 receiving placebo everyday for 14 days.
  Interventions: Drug: Leucettinib-21

INTERVENTIONS:
Drug: Leucettinib-21 — See arm's description.

SUMMARY:
Leucettinib-21 First-in-Human Phase 1 Study in 6 Parts: Single (Part 1 and 5) and Multiple (Part 3 and 6) Ascending Doses, and Food-Effect (Part 2) in Healthy Subjects, and Single Dose (Part 4) in People with Down Syndrome (DS) and Alzheimer's Disease (AD).

For Parts 1, 3, 4, 5 and 6, safety and tolerability of an oral administration of Leucettinib-21 will be assessed as primary objectives. Pharmacokinetics and pharmacodynamic biomarkers will be investigated as secondary objectives.

For Part 2, the effect of high fat meal will be evaluated on the pharmacokinetics parameters after an oral administration of Leucettinib-21.

ELIGIBILITY:
Inclusion criteria for Parts 1, 2, 3, 5 & 6:

* Part 5: Healthy male and female aged to 18-55 years inclusive / Part 6: Healthy male aged to 18-55 years inclusive
* Part 1, 2, 3, 5 & 6 for males: Must agree to adhere to the contraception requirements: use of condom by the male subject plus an effective method of contraception for the subject partner of childbearing potential from the time of informed consent signature up to 4 months after last IMP administration. Highly effective method of birth control such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intra uterine devices (IUDs), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle) / Part 5 for females of childbearing potential: Must agree to adhere to the contraception requirements: use for the subject of a highly effective method of birth control (defined as methods that can achieve a failure rate less than 1per 100 per year when used consistently and correctly) restricted to non-hormonal intra uterine device or non-hormonal intra uterine system, vasectomized partner and use of a second form of contraception. Hormonal methods of contraception whichever the mode of administration are not permitted. The following acceptable methods can be used as a second form of contraception during the study: partner's use of a condom or the subject's use of an occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam, gel, film, cream, or suppository from the time of informed consent signature and for 4 months after the last study drug administration. True sexual abstinence when this is in line with the preferred and usual lifestyle of the subject is acceptable. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of the trial and withdrawal are NOT acceptable methods of contraception / Part 5 for females of non-childbearing potential: female subjects who are postmenopausal (defined as spontaneous amenorrhea for at least 1 year or spontaneous amenorrhea for at least 6 months confirmed by follicle-stimulating hormone [FSH] result of ≥ 40 IU/mL) are eligible for this study and female subjects with surgical sterilization (i.e., bilateral tubal ligation/salpingectomy, hysterectomy) also;
* Non-smoker subject or smoker of not more than 5 cigarettes a day;
* Parts 1, 2, 3 & 6: Body Mass Index (BMI) between 18.5 and 28,0 (kg/m2) inclusive, with body weight between 60 and 100 kg inclusive, at Screening and Day -1 / Part 5: Body Mass Index (BMI) between 18.5 and 28,0 (kg/m2) inclusive, with body weight between 50 and 100 kg inclusive, at Screening and Day -1;
* Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
* Normal Blood Pressure (BP), oxygen saturation and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

  * 95 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg,
  * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
  * 45 bpm ≤ HR ≤ 90 bpm,
  * Or considered NCs by investigators;
* Normal ECG recording on a 12-lead ECG at the screening visit:

  * 120 ≤ PR < 210 ms,
  * QRS < 120 ms,
  * QTcf ≤ 430 ms for male,
  * No sign of any trouble of sinusal automatism,
  * Or considered NCs by investigators;
* Laboratory parameters within the normal range of the laboratory (hematology, hemostasis and blood biochemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non-relevant by the Investigator;
* Normal dietary habits;
* Signing a written informed consent prior to selection;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Non-inclusion criteria for Parts 1, 2, 3, 5 & 6:

* Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, infectious disease, endocrine, immunologic, dermatologic or/and any relevant disease;
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician;
* Symptomatic hypotension whatever the decrease of the blood pressure or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg or DBP equal to or greater than 10 mmHg within two minutes of changing from supine to standing position;
* Positive urine drug testing or alcohol testing at Screening or Day -1;
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests;
* Clinical symptoms suspected of acute infectious disease within 2 weeks before the first study drug administration;
* Any drug intake (except paracetamol) during the month prior to the first administration;
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day);
* Blood donation (including as part of a clinical trial) in the 2 months before administration;
* General anesthesia in the 3 months before administration;
* Inability to abstain from intense muscular effort;
* No possibility of contact in case of emergency;
* Excessive consumption of beverages with xanthine bases (>4cups or glasses/day);
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
* Persons deprived of their liberty by judicial or administrative decision; persons under coercive psychiatric care; adults under legal protection (guardianship/trusteeship); persons under court protection;
* Subject in the exclusion period of a previous study and within less than 4 weeks or 5 half-lives of the last administration of an experimental drug;
* Administrative or legal supervision;
* Subject who would receive more than 6000 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Main inclusion criteria for Part 4:

* Down Syndrome and Alzheimer's disease male individuals;
* Must agree to adhere to the contraception requirements;
* Non-smoker subject or smoker of not more than 5 cigarettes a day;
* Patient and/or their legal representatives (if applicable) are able to understand and provide written informed consent before starting any study-related activity according investigator judgment;
* Patient is able to participate fully in the study, be sufficiently proficient in the official language of the country in which they live, and be able to carry out study evaluations reliably;
* Blood Pressure (BP), oxygen saturation and Heart Rate (HR) at the screening visit after 10 minutes in supine position considered normal according the population or judged clinically non-relevant by investigators;
* ECG recording on a 12-lead ECG at the screening visit considered normal according the population or judged clinically non-relevant by investigators;
* Laboratory parameters within the normal range of the laboratory (hematology, hemostasis and blood biochemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non-relevant by the Investigator according the population;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research;
* Presence of an accompanying caregiver at the end of the study.

Main exclusion criteria for Part 4:

* Any relevant history or presence of significant diseases that would interfere with the assessment according the population except stabilized pathology with associated treatment for more than 3 months and known in the medical history;
* Patients considered unable to complete study assessments, according the investigator judgment;
* History of cancer in the past 5 years;
* History of inflammatory disease with potential for central nervous system involvement;
* Positive urine drug testing or alcohol testing at Screening or Day -1;
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Part 1 : Safety and tolerability of Leucettinib-21 after single administration at 6 increasing doses in healthy male subjects. | Part 1 : Up to 8 days following administration
  Assessment of systemic tolerability and safety
Part 2 : Effect of food on the PK parameters after an oral administration of Leucettinib-21 in healthy male subjects in high fat breakfast condition vs. under fasted conditions. | Part 2 : Up to 8 days following administration
  Plasma PK assessments
Part 3 : Safety and tolerability of Leucettinib-21 after multiple administration at 3 increasing doses in healthy male subjects | Part 3 : Up to 21 days following administration
  Assessment of systemic tolerability and safety
Part 4 : Safety and tolerability of Leucettinib-21 after single administration at 1 dose in Down Syndrome individuals and patients with Alzheimer's disease | Part 4 : Up to 8 days following administration
  Assessment of systemic tolerability and safety
Part 5 : Number of participants with treatment-related adverse events after single administration of Leucettinib-21 at 3 increasing doses in healthy male and female subjects. | Part 5 : Up to 8 days following administration
  Assessment of systemic tolerability and safety:
  * Adverse Events
  * Vital signs
  * Physical examination
  * ECG
  * Biological tests
Part 6 : Number of participants with treatment-related adverse events after repeated administration of Leucettinib-21 at 1 dose for 14 days in healthy male subjects | Part 6 : Up to 21 days following administration
  Assessment of systemic tolerability and safety:
  * Adverse Events
  * Vital signs
  * Physical examination
  * ECG
  * Biological tests
  * Psychometric tests (REST-SPER / FOCU SHIF)
  * Insulin, glucagon and somatostatin dosage
  * NT-pro BNP and troponin

SECONDARY OUTCOMES:
PK of Leucettinib-21 | Up to 24 hours following Leucettinib-21 administration
  Assessment of the plasmatic PK of Leucettinib-21
PD of Leucettinib-21 | Up to 4 hours following Leucettinib-21 administration
  Change in the proteome following Leucettinib-21 administration assessed by phosphoproteomics
Activity of DYRK1A | Up to 8 hours following Leucettinib-21 administration
  Change in DYRK1A activity following Leucettinib-21 administration assessed in Peripheral Blood Mononuclear Cells

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France